CLINICAL TRIAL: NCT03429842
Title: HIV Awal (Early) Testing & Treatment Indonesia Project Implementing 'Test and Treat' Strategies for HIV Treatment and Prevention in Key Populations in Indonesia: a Prospective Implementation Research Study (Phase 1 - Observational Phase)
Brief Title: HIV Awal (Early) Testing & Treatment Indonesia Project Observational Phase
Status: Completed | Type: Observational
Sponsor: Gadjah Mada University (Other)
Collaborators: World Health Organization (Other); Department of Foreign Affairs and Trade (DFAT), Australia (Unknown); Kirby Institute (Other Government); Hasan Sadikin General Hospital (Other); Sardjito Hospital Yogyakarta (Unknown); Yayasan Kerti Praja (Unknown); Udayana University (Other); Universitas Padjadjaran (Other); Universitas Katholik Atmajaya (Unknown)
Responsible Party: Principal Investigator, Prof. D N Wirawan, Prof. dr, MPH, Udayana University
Other Study IDs: The HATI Project HIV Phase 1
Record Dates: First submitted 2018-01-30; First posted 2018-02-12 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be one of the first to systematically evaluate strategies to improve the implementation of a T&T strategy in a concentrated epidemic in Asia.

While large controlled randomized trials assessing the efficacy of T&T at the community level are underway, they are being run in the generalised epidemic settings of Africa with the population HIV prevalence above 15%. Findings on implementation of T&T strategy from such settings will not be readily applicable to concentrated epidemics. This study will run in parallel with the trials so that the key implementation data in concentrated epidemic settings are available in a timely fashion. Finally, the study aims to develop capacity in implementation research in Indonesia.

In line with principles of implementation science, the components of the intervention package will be designed from extensive discussions with all stakeholders including affected communities. This will ensure that the intervention is acceptable, feasible and could be integrated in to larger policy framework beyond the study. Further, the study will utilize and explore the role of primary care centres (Puskesmas) in providing 'Test and Treat' services. The success of T&T strategy based on primary care model will be critical for the wider penetration of services to the key affected populations.

It will generate key data on critical steps in the cascade of care and show how current prevention services might enhance the uptake of HIV testing and immediate treatment. The study will identify which programmatic areas, under current resources, need strengthening for a larger scale implementation of T&T for HIV treatment and prevention.

This will be a prospective implementation research study assessing the impact of enhanced community based interventions, on the uptake of HIV treatment and retention in care among key populations as part of a T&T strategy in three urban settings in Indonesia. The enhanced package of interventions will be introduced in a series of steps over time.

This phase 1- Pre-implementation of the enhanced intervention package (Year 1) Current standard practices for HIV treatment and care will be observed ('business as usual'), utilising a comprehensive data collection system at each participating site. In accordance with current national guidelines, all HIV positive participants will be offered immediate ART initiation after being diagnosed as HIV positive.

DETAILED DESCRIPTION:
Purpose

The principal aims of the HATI study are:

1. To evaluate interventions aimed at increasing HIV testing and immediate antiretroviral therapy (ART), also known as the test and treat (T&T) strategy, in key populations in Indonesia;
2. To develop capacity in implementation research in Indonesia through training and the active participation of local researchers as investigators on the study.

The study will be conducted in two phases:

i) Phase 1 -observing current practice (year 1) ii) Phase 2 - after implementation of an enhanced intervention package (years 2 and 3)

Primary research objective

The primary objectives are to assess the impact of enhanced community based intervention compared with current practice, on:

1. Total number of virologically suppressed individuals from each key population (at the end of year 1 and year 4);
2. Proportion of people from each key population who are virologically suppressed 12 months after HIV diagnosis.

Analyses will be conducted separately for each key population

Secondary research objectives

1. To quantify and compare the HIV treatment cascade/continuum of care.
2. To assess safety of early ART and acceptability of early ART initiation.
3. To assess behavioural aspects of a T&T strategy, including impact on risk behaviours.

Research capacity building objectives

1. To enhance the capacity of senior local researchers as research leaders.
2. To increase the research skills and experience of early career researchers.

Study population

The study population will include adults from the following three key population groups:

i) Gay men and other men who have sex with men (MSM) ii) Female sex workers, including brothel and non-brothel based sex workers (FSW) iii) Waria (transgender people)

Study Design This will be a prospective implementation research study assessing the impact of enhanced community based interventions, on the uptake of HIV treatment and retention in care among key populations as part of a T&T strategy in three urban settings in Indonesia. The enhanced package of interventions will be introduced in a series of steps over time.

Phase 1- Pre-implementation of the enhanced intervention package (Year 1) Current standard practices for HIV treatment and care will be observed ('business as usual'), utilising a comprehensive data collection system at each participating site. In accordance with current national guidelines, all HIV positive participants will be offered immediate ART initiation after being diagnosed as HIV positive.

Phase2-a - Partial implementation of the enhanced package of interventions (Year 2) The components of an enhanced intervention package will be implemented selectively across the participating service delivery sites. The allocation of enhanced intervention package components across sites will be determined after the content of the package is developed in year 1 (see below for details describing how this package will be developed). Allocations will be made so as to allow for comparison between intervention and non-intervention exposure for each key population group.

Phase 2-b - Full implementation of the enhanced package of interventions (Years 3-4) The full implementation package will be implemented across all participating sites. Study outcomes for each phase will be compared. Participants will be followed up for a minimum of 12 months. The total study observation period will be 4 years.

In addition, during the first year of the study formative research will be conducted to inform the development of an enhanced package of interventions to increase the uptake of HIV testing and treatment, improved treatment adherence and treatment outcomes (virological suppression). This formative research will include focus group discussions and interviews with people from key populations, service providers, and other key stakeholders. The enhanced package will be designed such that it is locally relevant, acceptable to affected communities and deemed likely to be sustainable beyond the study by stakeholders.

Study sites The study will be undertaken in three urban locations in Bali, West Java and Yogyakarta. At each location a service providing HIV treatment will be designated as the Primary (Principal) Site; each Primary Site will be affiliated with a tertiary academic institution and will be responsible for overseeing the study activities in that location. A number of Satellite Sites will also be included in the study and will be involved in participant recruitment and/or follow-up.

Recruitment of HIV positive participants and sample size Eligible HIV positive individuals will be invited to enter the study following a positive HIV test during Phase 1 (year 1) and Phase 2 (years 2 and 3). The target total sample size across all three locations is 600 HIV positive MSM and 600 HIV positive FSW, with the aim to recruit, on average, 200 individuals from each population in each year .

Due to the considerably smaller overall waria population size there will be no specified target for the HIV positive waria sample.

HIV positive MSM, FSW and waria will be recruited at all locations. It is anticipated that recruitment is likely to be slower in Phase 1 (year 1) when no strategies in addition to current practice will be implemented to increase HIV testing; it is also anticipated that certain locations may recruit greater or fewer participants from each key population group. HIVpositive participants will be followed for the duration of the HATI study as far as possible.

Data on HIV testing among key populations Individuals from key populations receiving HIV test at participating study sites during Years 1-3 and who are found to be HIV-negative will not be recruited to the cohort in this study. De-identified data HIV testing among people from key populations will be analysed in order to examine patters in HIV testing during the study period.

Participant procedures Phase 1 :In line with a government directive on HIV treatment for people from key populations, all HIV positive participants will be offered immediate access to ART irrespective of CD4 count,. Linkage to HIV treatment and care, clinical management (including diagnostics) will be conducted as per routine practice. Costs borne by patients will remain as per current practices with exception of CD4 testing, which will be provided to study participants at no cost to them. Viral load testing at the time of being offered or starting treatment and every six months thereafter at no cost to the participant. Resistance testing will be done on virological failure, at no cost to the participant. A short behavioural questionnaire will be administered to all HIV positive participants at entry to the study and then every 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosis HIV Positive individual during the study observation period
* Aged 16 years and over
* Fow FSW : Had sex in exhange for money or a gft in the last 12 months or
* For MSM : Ever had sex with a man/waria
* For Waria : Identify as waria.

Exclusion criteria for all participants

* Unable to provide informed consent to enroll in the study
* Attending clinician judges that participation in the study would adversely affect individual.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include adults from the following three key population groups:
  i) Gay men and other men who have sex with men (MSM) ii) Female sex workers, including brothel and non-brothel based sex workers (FSW) iii) Waria (transgender people)
Sampling Method: Non-Probability Sample
Enrollment: 2071 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Rates of virological suppression under current practice | 12 months
  Number of participants viral load less than 50 copies/ml

SECONDARY OUTCOMES:
Uptake of HIV testing | 24 months
  Number of participants tested for HIV
Linkage between HIV testing and care | 24 months
  Number of HIV Positive participants registered with HIV care provider
Uptake of ART among FSW, MSM and waria | 24 months
  Number of HIV Positive Participants starting ART
Retention in treatment | 12 months
  Number of HIV Positive Participants retained in treatment after starting ART

CONTACTS AND LOCATIONS:
Overall Officials: Dewa N Wirawan, Prof, Principal Investigator — Universitas Udayana

REFERENCES:
- [Background] Januraga PP, Wulandari LP, Muliawan P, Sawitri S, Causer L, Wirawan DN, Kaldor JM. Sharply rising prevalence of HIV infection in Bali: a critical assessment of the surveillance data. Int J STD AIDS. 2013 Aug;24(8):633-7. doi: 10.1177/0956462413477556. Epub 2013 Jul 19. PMID 23970574
- [Background] Kotaki T, Khairunisa SQ, Sukartiningrum SD, Arfijanto MV, Utsumi T, Normalina I, Handajani R, Widiyanti P, Rusli M, Rahayu RP, Lusida MI, Hayashi Y, Nasronudin, Kameoka M. High prevalence of HIV-1 CRF01_AE viruses among female commercial sex workers residing in Surabaya, Indonesia. PLoS One. 2013 Dec 18;8(12):e82645. doi: 10.1371/journal.pone.0082645. eCollection 2013. PMID 24367533
- [Background] Safika I, Johnson TP, Cho YI, Praptoraharjo I. Condom Use Among Men Who Have Sex With Men and Male-to-Female Transgenders in Jakarta, Indonesia. Am J Mens Health. 2014 Jul;8(4):278-88. doi: 10.1177/1557988313508430. Epub 2013 Nov 7. PMID 24203992
- [Background] Mugglin C, Althoff NK, Wools-Kaloustian K, et al. Immunodeficiency at start of ART: A global view. 19th Conference on Retroviruses and Opportunistic Infections; 2012; Seattle, USA
- [Background] Karim SS, Karim QA. Antiretroviral prophylaxis: a defining moment in HIV control. Lancet. 2011 Dec 17;378(9809):e23-5. doi: 10.1016/S0140-6736(11)61136-7. Epub 2011 Jul 21. No abstract available. PMID 21771566
- [Background] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Mehendale S, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Wang L, Makhema J, Mills LA, de Bruyn G, Sanne I, Eron J, Gallant J, Havlir D, Swindells S, Ribaudo H, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano D, Essex M, Fleming TR; HPTN 052 Study Team. Prevention of HIV-1 infection with early antiretroviral therapy. N Engl J Med. 2011 Aug 11;365(6):493-505. doi: 10.1056/NEJMoa1105243. Epub 2011 Jul 18. PMID 21767103
- [Background] Granich RM, Gilks CF, Dye C, De Cock KM, Williams BG. Universal voluntary HIV testing with immediate antiretroviral therapy as a strategy for elimination of HIV transmission: a mathematical model. Lancet. 2009 Jan 3;373(9657):48-57. doi: 10.1016/S0140-6736(08)61697-9. Epub 2008 Nov 27. PMID 19038438
- [Background] Kato M, Granich R, Bui DD, Tran HV, Nadol P, Jacka D, Sabin K, Suthar AB, Mesquita F, Lo YR, Williams B. The potential impact of expanding antiretroviral therapy and combination prevention in Vietnam: towards elimination of HIV transmission. J Acquir Immune Defic Syndr. 2013 Aug 15;63(5):e142-9. doi: 10.1097/QAI.0b013e31829b535b. PMID 23714739
- [Background] Eaton JW, Johnson LF, Salomon JA, Barnighausen T, Bendavid E, Bershteyn A, Bloom DE, Cambiano V, Fraser C, Hontelez JA, Humair S, Klein DJ, Long EF, Phillips AN, Pretorius C, Stover J, Wenger EA, Williams BG, Hallett TB. HIV treatment as prevention: systematic comparison of mathematical models of the potential impact of antiretroviral therapy on HIV incidence in South Africa. PLoS Med. 2012;9(7):e1001245. doi: 10.1371/journal.pmed.1001245. Epub 2012 Jul 10. PMID 22802730
- [Background] Severe P, Juste MA, Ambroise A, Eliacin L, Marchand C, Apollon S, Edwards A, Bang H, Nicotera J, Godfrey C, Gulick RM, Johnson WD Jr, Pape JW, Fitzgerald DW. Early versus standard antiretroviral therapy for HIV-infected adults in Haiti. N Engl J Med. 2010 Jul 15;363(3):257-65. doi: 10.1056/NEJMoa0910370. PMID 20647201
- [Background] Kitahata MM, Gange SJ, Abraham AG, Merriman B, Saag MS, Justice AC, Hogg RS, Deeks SG, Eron JJ, Brooks JT, Rourke SB, Gill MJ, Bosch RJ, Martin JN, Klein MB, Jacobson LP, Rodriguez B, Sterling TR, Kirk GD, Napravnik S, Rachlis AR, Calzavara LM, Horberg MA, Silverberg MJ, Gebo KA, Goedert JJ, Benson CA, Collier AC, Van Rompaey SE, Crane HM, McKaig RG, Lau B, Freeman AM, Moore RD; NA-ACCORD Investigators. Effect of early versus deferred antiretroviral therapy for HIV on survival. N Engl J Med. 2009 Apr 30;360(18):1815-26. doi: 10.1056/NEJMoa0807252. Epub 2009 Apr 1. PMID 19339714
- [Background] Lockman S, Sax P. Treatment-for-prevention: clinical considerations. Curr Opin HIV AIDS. 2012 Mar;7(2):131-9. doi: 10.1097/COH.0b013e32834fcf6b. PMID 22227588
- [Background] Writing Committee for the CASCADE Collaboration. Timing of HAART initiation and clinical outcomes in human immunodeficiency virus type 1 seroconverters. Arch Intern Med. 2011 Sep 26;171(17):1560-9. doi: 10.1001/archinternmed.2011.401. PMID 21949165
- [Background] When To Start Consortium; Sterne JA, May M, Costagliola D, de Wolf F, Phillips AN, Harris R, Funk MJ, Geskus RB, Gill J, Dabis F, Miro JM, Justice AC, Ledergerber B, Fatkenheuer G, Hogg RS, Monforte AD, Saag M, Smith C, Staszewski S, Egger M, Cole SR. Timing of initiation of antiretroviral therapy in AIDS-free HIV-1-infected patients: a collaborative analysis of 18 HIV cohort studies. Lancet. 2009 Apr 18;373(9672):1352-63. doi: 10.1016/S0140-6736(09)60612-7. Epub 2009 Apr 8. PMID 19361855
- [Background] Suthar AB, Lawn SD, del Amo J, Getahun H, Dye C, Sculier D, Sterling TR, Chaisson RE, Williams BG, Harries AD, Granich RM. Antiretroviral therapy for prevention of tuberculosis in adults with HIV: a systematic review and meta-analysis. PLoS Med. 2012;9(7):e1001270. doi: 10.1371/journal.pmed.1001270. Epub 2012 Jul 24. PMID 22911011
- [Background] Forsyth AD, Valdiserri RO. Reaping the prevention benefits of highly active antiretroviral treatment: policy implications of HIV Prevention Trials Network 052. Curr Opin HIV AIDS. 2012 Mar;7(2):111-6. doi: 10.1097/COH.0b013e32834fcff6. PMID 22227586
- [Background] Garnett GP, Becker S, Bertozzi S. Treatment as prevention: translating efficacy trial results to population effectiveness. Curr Opin HIV AIDS. 2012 Mar;7(2):157-63. doi: 10.1097/COH.0b013e3283504ab7. PMID 22258503
- [Background] Bendavid E, Brandeau ML, Wood R, Owens DK. Comparative effectiveness of HIV testing and treatment in highly endemic regions. Arch Intern Med. 2010 Aug 9;170(15):1347-54. doi: 10.1001/archinternmed.2010.249. PMID 20696960
- [Background] Gardner EM, McLees MP, Steiner JF, Del Rio C, Burman WJ. The spectrum of engagement in HIV care and its relevance to test-and-treat strategies for prevention of HIV infection. Clin Infect Dis. 2011 Mar 15;52(6):793-800. doi: 10.1093/cid/ciq243. PMID 21367734
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Background] Uy J, Armon C, Buchacz K, Wood K, Brooks JT; HOPS Investigators. Initiation of HAART at higher CD4 cell counts is associated with a lower frequency of antiretroviral drug resistance mutations at virologic failure. J Acquir Immune Defic Syndr. 2009 Aug 1;51(4):450-3. doi: 10.1097/QAI.0b013e3181acb630. PMID 19474757
- [Background] Bastard M, Fall MB, Laniece I, Taverne B, Desclaux A, Ecochard R, Sow PS, Delaporte E, Etard JF. Revisiting long-term adherence to highly active antiretroviral therapy in Senegal using latent class analysis. J Acquir Immune Defic Syndr. 2011 May 1;57(1):55-61. doi: 10.1097/QAI.0b013e318211b43b. PMID 21775934
- [Background] Birger RB, Hallett TB, Sinha A, Grenfell BT, Hodder SL. Modeling the impact of interventions along the HIV continuum of care in Newark, New Jersey. Clin Infect Dis. 2014 Jan;58(2):274-84. doi: 10.1093/cid/cit687. Epub 2013 Oct 17. PMID 24140971
- [Background] Peters DH, Adam T, Alonge O, Agyepong IA, Tran N. Implementation research: what it is and how to do it. BMJ. 2013 Nov 20;347:f6753. doi: 10.1136/bmj.f6753. No abstract available. PMID 24259324
- [Background] Padian NS, Holmes CB, McCoy SI, Lyerla R, Bouey PD, Goosby EP. Implementation science for the US President's Emergency Plan for AIDS Relief (PEPFAR). J Acquir Immune Defic Syndr. 2011 Mar 1;56(3):199-203. doi: 10.1097/QAI.0b013e31820bb448. No abstract available. PMID 21239991
- [Background] Sohn AH, Srikantiah P, Sungkanuparph S, Zhang F. Transmitted HIV drug resistance in Asia. Curr Opin HIV AIDS. 2013 Jan;8(1):27-33. doi: 10.1097/COH.0b013e32835b804f. PMID 23196932
- [Derived] Widyanthini DN, Januraga PP, Wisaksana R, Subronto YW, Sukmaningrum E, Kusmayanti NA, Dewi H, Law M, Kaldor JM, Wirawan DN. HIV self-testing for men who have sex with men: an implementation trial in Indonesia. AIDS Care. 2022 Apr;34(4):527-534. doi: 10.1080/09540121.2021.1883509. Epub 2021 Feb 8. PMID 33550846
- [Derived] Januraga PP, Reekie J, Mulyani T, Lestari BW, Iskandar S, Wisaksana R, Kusmayanti NA, Subronto YW, Widyanthini DN, Wirawan DN, Wongso LV, Sudewo AG, Sukmaningrum E, Nisa T, Prabowo BR, Law M, Cooper DA, Kaldor JM. The cascade of HIV care among key populations in Indonesia: a prospective cohort study. Lancet HIV. 2018 Oct;5(10):e560-e568. doi: 10.1016/S2352-3018(18)30148-6. Epub 2018 Aug 22. PMID 30143455
- See also: UNAIDS. UNAIDS Report on the global AIDS epidemic. 2012 — http://www.unaids.org/en/media/unaids/contentassets/documents/epidemiology/2012/gr2012/20121120_UNAIDS_Global_Report_2012_with_annexes_en.pdf
- See also: UNAIDS. HIV in Asia and the Pacific:Getting to zero. 2011 — http://www.unaids.org/en/media/unaids/contentassets/documents/unaidspublication/2011/20110826_APGettingToZero_en.pdf
- See also: World Health Organization (WHO). Antiretroviral Treatment as Prevention (TasP) of HIV and TB. 2012 — http://whqlibdoc.who.int/hq/2012/WHO_HIV_2012.12_eng.pdf
- See also: UNAIDS. Indonesia's Minister of Health promises to transform the national response to AIDS. 2012 — http://www.unaids.org/en/resources/presscentre/featurestories/2012/october/20121023indonesia/